CLINICAL TRIAL: NCT03195101
Title: Evaluation of Transconjunctival Approach in Management of Orbital Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Abdelnasser Awad, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200091
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Orbital Tumors
Keywords: orbital tumors; transconjunctival approach

STUDY DESIGN:
Intervention Model Description: Incisional or excisional biopsy of orbital tumors via transconjunctival approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with orbital tumors (Experimental): patients with orbital tumors will be managed by excisional or incisional biopsy via the transconjunctival orbitotomy approach
  Interventions: Procedure: transconjunctival orbitotomy approach

INTERVENTIONS:
Procedure: transconjunctival orbitotomy approach — approach the orbital tumor through an incision in the conjunctiva, This is followed by blunt dissection of the tenons capsule. A traction suture is applied over the corresponding rectus muscle to guide the globe toward the desired direction. The orbital fat is retracted by malleable retractor and blunt dissection through the orbital connective tissue continues until reaching the edge of the tumor. After the mass is exposed, a biopsy or complete resection of the mass is taken place

SUMMARY:
Many surgical approaches for excision of orbital tumors have been described. These approaches do not allow access to all orbital quadrants. Furthermore, some of these approaches are technically difficult, associated with long morbidity and post operative pain, having high rate of complications or having unacceptable cosmetic appearance. the investigators present the transconjunctival approach as an alternative procedure that allows access to orbital tumors in different locations as well as less morbidity and better cosmetic results

DETAILED DESCRIPTION:
Orbital tumors are divided anatomically into intraconal and extraconal depending on their relationship with the muscle cone which is further classified into anterior and posterior orbital tumors. Excision of orbital tumors is considered a challenge for the surgeon. This is due to the complex structure of the orbit. The orbital cavity is narrow that does not allow adequate exposure. Furthermore, the orbit is full of vital structures which require careful manipulation. Many surgical approaches for excision of these tumors have been described. These approaches do not allow access to all orbital quadrants. Furthermore, some of these approaches are technically difficult, associated with long morbidity and post operative pain due to the osteotomy, having high rate of complications or having unacceptable cosmetic appearance. Few studies with limited number of patients have used transconjunctival approach in management of orbital tumors All patients with orbital tumor will be managed by the transconjunctival incisional or excisional biopsy according to the suggested nature of the tumor being benign or malignant as well as the site of the tumor using the clinicoradiological finding. In case of intraconal tumors, the mass will be approached via the transconjunctival approach but if the mass is out of reach via this approach, lateral orbitotomy approach will be used as an alternative procedure to perform the predetermined decision. This allows detection of the intraconal tumor criteria that could be excised safely via this approach

ELIGIBILITY:
Inclusion Criteria:

* Patients with orbital tumor either benign or malignant.

Exclusion Criteria:

* Patients with apical tumors not accessible with transconjunctival approach.
* Patients with too anterior tumors (superficial dermoid and lacrimal gland swelling).
* Patients with non-neoplastic orbital lesions.
* Patients with follow up period of less than 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
successfulness of the surgical procedure | every patient will be assessed 3 days postoperative
  The procedure will be considered successful if the predetermined decision is achieved without sight threatening complications. The procedure will be considered a failure if the decision could not be achieved or if a sight threatening complication occurs.

SECONDARY OUTCOMES:
Early and late complications of the approach and their long term effects | 3 days postoperative, 1 week, 1 month and 3 months postoperative.
  the assessment will include intraoperative or postoperative complications. the complication will be followed up for up to three months to determine if the complication is self limited (example: self limited lid edema or subconjunctival hemorrhage) or has a long term effect (example: permanent visual loss or permanent limited ocular motility)

IPD SHARING:
Plan to Share IPD: No